CLINICAL TRIAL: NCT07393750
Title: High-Power Laser Versus Pulsed Eectromagnetic Therapy on Pain and Hoffman Reflex in Lumbar Radiculopathy.
Brief Title: High-power Laser Versus Pulsed Electromagnetic Therapy in Lumbar Radiculopathy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Menna Tallah Sherif Hassan, Physiotherapist Egyptair Hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006166
Record Dates: First submitted 2026-01-24; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Radiculopathy; Hoffman's Reflex; Pulsed Electromagnetic Therapy; Laser Therapy; Herniated Lumbar Disc
MeSH Terms: conditions — Radiculopathy; Reflex, Abnormal

STUDY DESIGN:
Intervention Model Description: Randomized Control Study The selected patients will be randomly assigned into "three" equal groups: study group 1 (G1a), study group 2 (G1b) and control group (G2). The control group patients will receive selected physiotherapy program. The study group (G1a) will receive 20 minutes of high-power laser therapy followed by 25 the same physical therapy program as control group. The study group 2 patients will receive 20 minutes of Pulsed electromagnetic field followed by 25 the same selected physiotherapy program as control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study group 1 (G1a) (Experimental): study group (G1a) will receive 20 minutes of high-power laser therapy followed by 25 the same physical therapy program as control group.
  Interventions: Device: high-power laser; Other: physiotherapy program
- study group 2 (G1b) (Experimental): The study group 2 patients will receive 20 minutes of Pulsed electromagnetic field followed by 25 the same selected physiotherapy program as control group.
  Interventions: Device: Pulsed electromagnetic field; Other: physiotherapy program
- control group (G2) (Experimental): The control group patients will receive selected physiotherapy program.
  Interventions: Other: physiotherapy program

INTERVENTIONS:
Device: high-power laser — The study group (G1a) receive 20 minutes of high-power laser therapy followed by 25 the same physical therapy program as control group.
  Arms: study group 1 (G1a)
Device: Pulsed electromagnetic field — group 2 patients will receive 20 minutes of Pulsed electromagnetic field followed by 25 the same selected physiotherapy program as control group.
  Arms: study group 2 (G1b)
Other: physiotherapy program — Selected Physical therapy program in the form of:
  1. Nerve gliding exercise for sciatic nerve.
  2. Hot pack for 15 minutes, for 12 sessions.
  3. Core stability exercise (static abdominal exercise, bridging, knee to chest).

SUMMARY:
To compare between high-power laser versus pulsed electromagnetic therapy on pain and Hoffman reflex in lumbar radiculopathy.

DETAILED DESCRIPTION:
Lumbar radiculopathy is one of the most common complaints evaluated by a spine surgeon. Its prevalence has been estimated to be 3%-5% of the population, affecting both men and women. Age is a primary risk factor, as it occurs secondary to the degenerative process within the spinal column. Symptoms typically begin in midlife, with men often affected in the 40s while women are affected in the 50s and 60s. Disc herniation is one of the primary causes of lumbar radiculopathy.

The pressure exerted by the herniated disc on the longitudinal ligament and the local inflammation results in localized back pain. The lumbar radicular pain arises when disc material exerts pressure or contacts the thecal sac or lumbar nerve roots, resulting in nerve root ischemia and inflammation. The annulus fibrosus is thinner on the posterolateral aspect and lacks support from the posterior longitudinal ligament, making it vulnerable to herniations. Due to the proximity of the nerve root, a posterolateral herniation is more likely to result in nerve root compression.

High Intensity Power Laser (HILT) delivers high-intensity light energy to deep tissues in short pulses (120-200 µs). It causes minor and slow light absorption by the chromophores, which increases mitochondrial bioenergetics by causing extra adenosine triphosphate synthesis and oxygen consumption, as well as RNA and DNA production, resulting in tissue stimulation. Various studies have shown that laser light has anti-inflammatory and analgesic effects and that it reduces edema. HILT also has photothermal properties, resulting from the transformation of high-energy light into heat in tissue.

Magnetic therapy is considered as a safe, easy and non-invasive physical therapy modality used to treat pain, inflammation and other types of pathologies and diseases. Pulsed electromagnetic field (PEMF) refers to a basic law of electromagnetism that describes how a magnetic field interacts with an electric circuit to produce an electromotive force known as electromagnetic induction. Exposure to PEMF has been reported to modulate neuronal excitation and neurogenesis related to Na+ channel activity. Neurons excited by the exogenous electromagnetic force can also affect neighboring cells by ephaptic interaction. They also modulate levels of various growth factors that prevent autoimmune disease and inhibit tissue degeneration.

The H-reflex or "Hoffmann reflex" is obtained by electrode stimulation of the posterior tibial nerve in the popliteal space-at a slow rate with long duration-submaximal electrical shock, and recorded with surface electrodes over the gastrocnemius-soleus complex. The impulse travels up the sensory fibers to the spinal cord, synapses with the alpha motor neuron and returns down the motor fibers to the calf muscle. H-reflex latencies are long, in the 40 to 45 msec range. They are mostly carried out in the S1 root distribution and cannot be recorded consistently from other muscles.

Statement of the problem Is there any difference between high-power laser versus pulsed electromagnetic therapy on pain and hoffman reflex in lumbar radiculopathy?

Purposes of the study:

To compare between high-power laser versus pulsed electromagnetic therapy on pain and Hoffman reflex in lumbar radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* • Sixty lumbar radiculopathy patients, of both sexes, will represent the sample.

  * The patient's age will range from 55 to 68 years old.
  * Patients with degenerative lumbar disc lesion at L5-S1 confirmed by MRI and latency in H- reflex.
  * Patients with unilateral sciatic radiating pain (from 5 to 8 by visual analogue scale).
  * Patient with normal cognitive function (MME more than 25)
  * BMI from 20-29.9

Exclusion Criteria:

* The patients will be excluded if they have one of the followings:

  1. Patients with pacemakers and presence of electronic implants.
  2. Pregnant women.
  3. History of or existing malignant conditions, active tuberculosis of the lungs.
  4. Any medical condition that may cause sciatic nerve lesion except lumbar radiculopathy, (e.g., diabetes mellitus or collagen disorders).
  5. Cardiac, renal or hepatic failures recent or previous history of seizures or epilepsy.
  6. Previous surgery at L5-S1.
  7. Bleeding disorders.
  8. Serious infections of a viral, bacterial and fungal origin, conditions after organ transplants, upper motor neuron lesions.
  9. Patients with cognitive impairment.

Ages: 55 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-29 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | baseline
  The Visual Analogue Scale (VAS) is a tool for measuring pain intensity, using a continuous 10-centimeter line with "no pain" at one end (0) and "worst imaginable pain" at the other (10), where patients mark their current pain level, with a ruler used to measure the score from the zero mark for a score out of 10, commonly used in research and clinical settings to track pain changes.
Hoffman reflex or H reflex | baseline
  H-reflex will be measured in the soleus muscle by stimulating the tibial nerve with a one-millisecond pulse at 0.2pps of H-max. The peak-to-peak amplitude of the highest recorded H-reflex and the latencies of four spaced traces for both lower extremities will be averaged for each participant. The soleus H-reflex will be evoked by tibial nerve stimulation in the popliteal fossa.

CONTACTS AND LOCATIONS:
Overall Officials: PROF. DR. MOSHERA HASSAN DARWISH, Professor of Physical Therapy, Study Chair — Cairo University
Locations (1):
- Egyptair Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/b978-0-444-64032-1.00014-x
- See also: Related Info — https://doi.org/10.1016/j.anclin.2011.04.004
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK482431/
- See also: Related Info — https://doi.org/10.1007/s00586-024-08528-8
- See also: Related Info — https://doi.org/10.1016/j.clinph.2010.03.004
- See also: Related Info — https://doi.org/10.1186/s13244-023-01514-6
- See also: Related Info — https://doi.org/10.1016/b978-0-12-385157-4.00689-8
- See also: Related Info — https://www.hopkinsmedicine.org/health/conditions-and-diseases/lumbar-disc-disease-herniated-disc
- See also: Related Info — https://emedicine.medscape.com/article/95025-overview
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK560878/
- See also: Related Info — https://doi.org/10.21873/invivo.12300
- See also: Related Info — https://doi.org/10.12680/balneo.2023.594
- See also: Related Info — https://doi.org/10.1016/j.mehy.2024.111485